CLINICAL TRIAL: NCT02924831
Title: High-tech Acupuncture for Treatment of Chronic Fatigue Syndrome - A Sino-Austrian Cooperation Randomized Controlled Trial(RCT) on Heart Rate Variability
Brief Title: High-tech Acupuncture for Treatment of Chronic Fatigue Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hubei Provincial Collaborative Innovation Center of Preventive Treatment by Acupuncture and Moxibust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XTCX2016-QXZ
Record Dates: First submitted 2016-09-27; First posted 2016-10-05 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-07

CONDITIONS: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Acupuncture Therapy; Moxibustion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Moxibustion group (Experimental): drug:moxa Moxibustion was to stimulate acupoints of Guanyuan(RN4)and the Zusanli(ST36) with burned moxa.
  Interventions: Other: moxibustion
- Acupuncture group (Experimental): material: stainless steel needle In acupuncture treatment, needles were applied to acupoints of Guanyuan(RN4)and Zusanli(ST36),with manipulations to get Deqi sensation.
  Interventions: Other: Acupuncture
- Placebo group (Placebo Comparator): material: stainless steel needle Needles were applied to acupoints of Guanyuan(RN4)and Zusanli(ST36),but without any manipulations and Deqi sensation.
  Interventions: Other: placebo
- Zusanli（ST36)-acupuncture group (Experimental): material: stainless steel needle Stimulating acupoints of Zusanli(ST36) with acupuncture.
  Interventions: Other: Acupuncture
- Guanyuan(RN4)-acupuncture group (Experimental): material: stainless steel needle. Stimulating acupoint of Guanyuan(RN4) with acupuncture.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Stimulating acupoints by using stainless steel needles with manual manipulation.
  Arms: Acupuncture group; Guanyuan(RN4)-acupuncture group; Zusanli（ST36)-acupuncture group
Other: moxibustion — Stimulating acupoints by using burned moxa
  Arms: Moxibustion group
Other: placebo — Stimulating acupoints by using stainless steel needles without manual manipulation.
  Arms: Placebo group

SUMMARY:
1. To study the relationship between Chronic Fatigue Syndrome (CFS) and heart rate (HR) and its variability (HRV).
2. To compare the curative effects and the HR/HRV indices between applicationa of different acupoints as well as different treatments (acupuncture and moxibustion).

ELIGIBILITY:
Inclusion Criteria:

1. The patients meeting criteria of CFS;
2. Aged from 18-65;
3. With no skin lesions for the acupuncture area;
4. Sign on the Informed Consent Form;

Exclusion Criteria:

1. Patients who can't accept and are afraid of acupuncture in the acupuncture group.
2. Patients suffering from heart and cerebrovascular diseases, serious lung disease, diabetes, neurological diseases, or severe primary diseases such as those of liver, kidney and the hematopoietic system.
3. Persons suffering from a mental disease, Alzheimer's disease or cancer.
4. Persons who have taken qi-reinforcing Chinese herbal medicine in the week preceding the investigation.
5. Pregnant women and nursing mothers.
6. Persons suffering from thrombocytopenia and abnormalities of blood coagulation function.
7. Persons with alcohol and drug abuse history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-05 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Chalder's Fatigue Scale Score(CFSS) | Two years
  In CFSS, symptoms of fatigue are assessed by scores ranging from 0 to 3.

SECONDARY OUTCOMES:
Numeric Rating Scale(NRS) | Two years
  NRC is a 10cm scale to assess the fatigue degree ranging from 0 to 10, the score of 0 stands for 'no fatigue' and 10 for 'serious'.
36-item Short-Form Health Survey (SF-36) | Two years
  SF-36 consists of 36 items categorized as 8 dimensions: social functioning (2 items), role limitation-emotion (3 items), mental health (5 items), physical functioning (10 items), role limitation-physical (4 items), bodily pain (2 items), vitality (4 items), general health (5 items) and 1 question of health change in recent one year.
Deficiency of Qi Scale Score (DQSS) | Two years
  In DQSS, symptoms are assessed by scores ranging from 1 to 3, which stand for 'mild' to 'serious'.
Total Power(TP) | Two years
  Total Power of heart rate variability(HRV) (ms²/Hz, %)), detected by portable HRV device.
Low frequency(LF) | Two years
  Low frequency band (ms²/Hz, %), detected by portable HRV device.
High frequency (HF) | Two years
  High frequency band (ms²/Hz, %), detected by portable HRV device.
LF/HF | Two years
  Ratio of LF and HF frequency band powers (ms²/Hz, %), calculated by LF and HF results.
Ultra-low frequency(ULF) | Two years
  Ultra-low frequency band (ms²/Hz, %),detected by portable HRV device.
Very low frequency | Two years
  Very low frequency band (ms²/Hz, %),,detected by portable HRV device.

CONTACTS AND LOCATIONS:
Locations (1):
- Hubei university of TCM, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li T, Litscher G, Zhou Y, Song Y, Shu Q, Chen L, Huang Q, Wang Y, Tian H, Teng R, Wang H, Liang F. Effects of acupuncture and moxibustion on heart rate variability in chronic fatigue syndrome patients: Regulating the autonomic nervous system in a clinical randomized controlled trial. Complement Ther Med. 2025 Sep;92:103184. doi: 10.1016/j.ctim.2025.103184. Epub 2025 Apr 30. PMID 40315935